CLINICAL TRIAL: NCT04018144
Title: PPAR-γ, RXR-α, and VDR Expressions in Periodontitis Patients With Different Stage and Grade Involvement
Brief Title: Running Title: PPAR-γ, RXR-α, and VDR Expressions in Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Özkan Karataş, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: Gaziosmanpasa University Per
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis
Keywords: Periodontitis, PPAR-γ, RXR-α, VDR
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group-1: Healthy individuals
  Interventions: Diagnostic Test: Gingiva Biopsy Sampling
- Group-2: Periodontitis patients-stage 3-grade B
  Interventions: Diagnostic Test: Gingiva Biopsy Sampling
- Group-3: Periodontitis patients-stage 3-grade C
  Interventions: Diagnostic Test: Gingiva Biopsy Sampling

INTERVENTIONS:
Diagnostic Test: Gingiva Biopsy Sampling — Gingival samples of healthy individuals were collected by gingivectomy or crown lengthening procedure in the routine treatment protocol or before orthodontically indicated tooth extraction. Gingival samples of periodontitis patients were obtained during the scaling and root planning procedure. Posterior maxillary teeth (#4, #5, #6, and #7) were chosen for gingival sampling.

SUMMARY:
Objective: The present study aimed to determine the expressions of nuclear receptors PPAR (Peroxisome proliferative activator receptor)-γ, RXR (Retinoid X receptor)-α, and vitamin D receptor (VDR) in healthy volunteers and periodontitis patients with different grade involvement.

Methods: Group-1; healthy individuals, Group-2; periodontitis patients-stage 3 grade B, (H-GradeB), Group-3; periodontitis patients-stage 3 grade C, (D-GradeC). Clinical parameters as plaque index (PI), gingival index (GI) and clinical attachment levels (CAL) were measured. Fibroblast and inflammatory cells, PPAR-γ, RXR-α, and VDR levels were determined in histological slides.

ELIGIBILITY:
Inclusion Criteria:

* systemic health
* no drug use
* no previous periodontal treatment within six months
* no tobacco use

Exclusion Criteria:

* pregnant or lactating women
* patients used antibiotics in the last 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three study groups were created, and 45 participants were enrolled in the present study.
  The study groups were; Group-1; healthy individuals (mean age 42.34±3.89, nine women, six men) Group-2; periodontitis patients-stage 3 grade B, (GradeB) (mean age 43.12±3.16, 10 women, 5 men) Group-3; periodontitis patients-stage 3 grade C, (GradeC) (mean age 42.78±2.99, 10 women, 5 men)
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cell counts | During histological tissue processing
  Connective tissues were evaluated, and inflammatory cell infiltration were counted in the H&E stained slides using a light microscope (Nikon Eclipse, E 600, Tokyo, Japan). For cell counting, connective tissue neighboring gingival epithelium was marked, and a cell counting frame of 10000 µm2 was marked. Inflammatory cells (neutrophil, lymphocyte, eosinophil, and macrophage cells) within the frame were counted. The measurements were performed from three different points, and the mean of these three measurements was recorded.
Fibroblasts counts | During histological tissue processing
  For cell counting, connective tissue neighboring gingival epithelium was marked, and a cell counting frame of 10000 µm2 was marked. The fibroblast counts within the frame were counted. The measurements were performed from three different points, and the mean of these three measurements was recorded.
PPAR (Peroxisome proliferative activator receptor)-γ | During histological tissue processing
  PPAR (Peroxisome proliferative activator receptor)-γ levels were determined via immunohistochemistry.
RXR (Retinoid X receptor)-α | During histological tissue processing
  RXR (Retinoid X receptor)-α levels were determined via immunohistochemistry.
Vitamin D receptor (VDR) | During histological tissue processing
  Vitamin D receptor (VDR) levels were determined via immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No